CLINICAL TRIAL: NCT04317664
Title: Intervention to Improve Driving Practices Among High-Risk Teen Drivers
Acronym: projectDRIVE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ginger Yang (Other)
Collaborators: University of Iowa (Other); Ohio State University (Other); University of Nebraska (Other)
Responsible Party: Sponsor-Investigator, Ginger Yang, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1
Record Dates: First submitted 2020-03-04; First posted 2020-03-23 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Drive; Recidivism; Communication; Feedback, Psychological
MeSH Terms: conditions — Recidivism; Communication | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Control Group (No Intervention): The Control Group will have the in-vehicle device installed in the teen's car, but all feedback features will be disabled.
- Feedback Only Group (Experimental): The Feedback Only Group will have the in-vehicle devices in the teen's car and download the smartphone app on the teen's smartphone. Researchers will provide instructions on how teens can review their driving data. Teens will also receive biweekly cumulative driving reports.
  Interventions: Combination Product: In-vehicle device
- Feedback and Parent Communication Group (Experimental): The Feedback and Parent Communication Group will have the in-vehicle devices in the teen's car and download the smartphone app on the teen's smartphone. Researchers will provide instructions on how teens and parents can review their driving data. The parent will also receive communication training on how to motivate their teen to adopt safe driving habits via online modules and a video call with a motivational interviewing professional. A second booster session will also occur two months after the initial training. Both teens and parents will receive a biweekly cumulative driving report.
  Interventions: Combination Product: In-vehicle device; Behavioral: Parent Communication

INTERVENTIONS:
Combination Product: In-vehicle device — The Azūga™ in-vehicle driving feedback technology, which consists of a pager-sized device plugged into the vehicle's on-board diagnostic port (installed in the teen's car) and a smartphone app (downloaded on the teen's smartphone), will be installed/downloaded. Three types of feedback will be provided to intervention teens: 1) Direct audio feedback from the installed device; 2) Detailed cumulative driving data; and 3) A customized biweekly driving summary report.
  Other Names: Azuga device; OBDII device; In-vehicle Driving Feedback Technology
  Arms: Feedback Only Group; Feedback and Parent Communication Group
Behavioral: Parent Communication — An individualized virtual training in communication strategies about driving safety along with a booster session will be delivered by a traffic safety communication specialist to subjects in the Feedback and Parent Communication Group. Intervention parents in this group will also be provided with access to an online parent-teen safe driving communication guide.
  Other Names: Motivational Interviewing; Steering Teens Safe; Parent Training
  Arms: Feedback and Parent Communication Group

SUMMARY:
The purpose of this study is to test the effects of an in-vehicle driving feedback technology, with and without parent communication training, on risky driving events, unsafe driving behaviors, and subsequent traffic violations among teens who have recently received a moving traffic violation.

DETAILED DESCRIPTION:
For this study, 240 teen and parent/guardian dyads will be randomized into one of three study groups for six months. Teens will be aged 16-17 who committed a moving-related traffic violation and their parent/legal guardian who is most involved with their driving. Researchers will aim to determine the effects of the intervention on teens' risky driving events, unsafe driving behaviors, and traffic violation recidivism. Additionally, researchers will aim to determine the effects of the intervention on frequency and quality of parent-teen communications about safe driving practices.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-17 years at time of violation
* Convicted of a moving violation
* Possess a valid intermediate driver's license issued by the state of Ohio, with proof of car insurance
* Access to a vehicle with an On-board Diagnostics II system port (i.e. cars made after 1996) in which he/she is the primary driver
* Smartphone with Bluetooth capabilities
* At least one legal guardian

Exclusion Criteria:

* Unable to drive due to injury, license suspension, or car damage
* Vehicle already has an in-vehicle driving feedback system installed
* Extremely low average weekly drive time (e.g. <1 hour per week)
* Currently enrolled in another driving-related study
* War of the State
* Non-English speaking parent
* Adults unable to consent
* Pregnant women
* Prisoners

Ages: 16 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 480 (Estimated)
Dates: Start 2020-09-28 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Number of Risky Driving Events | Six months/study period
  Events of hard braking and sudden acceleration.
Number of Unsafe Driving Behaviors | Six months/study period
  Events of speeding, distracted driving, and no seatbelt use.
Frequency of Parent-teen Communication | Six months/study period
  Frequency of parent-teen communication about driving safety. This will be measured through a survey asking parents how often they discussed a driving topic with their teen.
Recidivism | Up to one year post-study period
  Recidivism will be measured among teens in all three groups by linking traffic citations and court disposition data with the participating teen's driver's license number. Recidivism during the 12 months following enrollment, including date and type of violation, and days from index violation to subsequent violation will be analyzed.
Quality of Parent-teen Communication | Six months/study period
  The quality of parent-teen communication about driving safety will be measured through an average rating of each driving topic which is recorded by the parent and teen.

OTHER OUTCOMES:
Engagement with Parent Communication Training | Six months/study period
  Engagement with the parent communication training will be measured among parents in the Feedback and Parent Communication Group using online measurements.
Engagement with Device Feedback | Six months/study period
  Engagement with device feedback will be measured among teens in the Feedback Only Group and the Feedback and Parent Communication Group and parents in the Feedback and Parent Communication Group via online tracking of the participant's web interface using Google Analytics.

CONTACTS AND LOCATIONS:
Overall Officials: Jingzhen (Ginger) Yang, PhD, MPH, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data used and/or analyzed during this study, along with detailed study protocol, are available from the PI, Dr. Jingzhen Yang, on reasonable request. The data are not publicly available due to privacy restrictions.
Supporting Information: Study Protocol, SAP
Time Frame: Starting 6 months after the summary data are published.
Access Criteria: De-identified data for the study and a data dictionary will be made available to other researchers following approval of a study proposal by the PI, Dr. Jingzhen Yang(ginger.yang@nationwidechildrens.org). The study protocol and statistical analysis plan are also available from the PI, Dr. Jingzhen Yang.

REFERENCES:
- [Background] Centers for Disease Control and Prevention. Data and Statistics (WISQARS). www.cdc.gov/injury/wisqars. Accessed February 1, 2016.
- [Background] Insurance Institute for Highway Safety (IIHS). Fatality facts: teenagers 2013. Arlington, VA: http://www.iihs.org/iihs/topics/t/teenagers/fatalityfacts/teenagers. Accessed February 1, 2016.
- [Background] Williams AF. Teenage drivers: patterns of risk. J Safety Res. 2003 Jan;34(1):5-15. doi: 10.1016/s0022-4375(02)00075-0. PMID 12535901
- [Background] Mayhew DR, Simpson HM, Pak A. Changes in collision rates among novice drivers during the first months of driving. Accid Anal Prev. 2003 Sep;35(5):683-91. doi: 10.1016/s0001-4575(02)00047-7. PMID 12850069
- [Background] McCartt AT, Shabanova VI, Leaf WA. Driving experience, crashes and traffic citations of teenage beginning drivers. Accid Anal Prev. 2003 May;35(3):311-20. doi: 10.1016/s0001-4575(02)00006-4. PMID 12643948
- [Background] Jonah BA, and Dawson NE. Youth and risk: age differences in risky driving, risk perception, and risk utility. Alcohol, Drugs and Driving. 1987;3(3):13-29.
- [Background] Summala H, Rajalin S, Radun I. Risky driving and recorded driving offences: a 24-year follow-up study. Accid Anal Prev. 2014 Dec;73:27-33. doi: 10.1016/j.aap.2014.08.008. Epub 2014 Aug 27. PMID 25171522
- [Background] Alver Y, Demirel MC, Mutlu MM. Interaction between socio-demographic characteristics: traffic rule violations and traffic crash history for young drivers. Accid Anal Prev. 2014 Nov;72:95-104. doi: 10.1016/j.aap.2014.06.015. Epub 2014 Jul 12. PMID 25019690
- [Background] Ayuso M, Guillen M, Alcaniz M. The impact of traffic violations on the estimated cost of traffic accidents with victims. Accid Anal Prev. 2010 Mar;42(2):709-17. doi: 10.1016/j.aap.2009.10.020. Epub 2009 Nov 22. PMID 20159098
- [Background] Factor R. The effect of traffic tickets on road traffic crashes. Accid Anal Prev. 2014 Mar;64:86-91. doi: 10.1016/j.aap.2013.11.010. Epub 2013 Dec 2. PMID 24342150
- [Background] Gebers MA, Peck RC. Using traffic conviction correlates to identify high accident-risk drivers. Accid Anal Prev. 2003 Nov;35(6):903-12. doi: 10.1016/s0001-4575(02)00098-2. PMID 12971925
- [Background] Goldenbeld C, Reurings M, Van Norden Y, Stipdonk H. Crash involvement of motor vehicles in relationship to the number and severity of traffic offenses. An exploratory analysis of Dutch traffic offenses and crash data. Traffic Inj Prev. 2013;14(6):584-91. doi: 10.1080/15389588.2012.743125. PMID 23859422
- [Background] Chen W, Cooper P, and Pinili M. Driver accident risk in relation to the penalty point system in British Columbia. J Safety Res. 1995;26:9-18.
- [Background] Cooper PJ. The relationship between speeding behaviour (as measured by violation convictions) and crash involvement. J Safety Res. 1997;28:83-95.
- [Background] Rajalin S. The connection between risky driving and involvement in fatal accidents. Accid Anal Prev. 1994 Oct;26(5):555-62. doi: 10.1016/0001-4575(94)90017-5. PMID 7999200
- [Background] Carney C, McGehee DV, Lee JD, Reyes ML, Raby M. Using an event-triggered video intervention system to expand the supervised learning of newly licensed adolescent drivers. Am J Public Health. 2010 Jun;100(6):1101-6. doi: 10.2105/AJPH.2009.165829. Epub 2010 Apr 15. PMID 20395588
- [Background] Farmer CM, Kirley BB, McCartt AT. Effects of in-vehicle monitoring on the driving behavior of teenagers. J Safety Res. 2010 Feb;41(1):39-45. doi: 10.1016/j.jsr.2009.12.002. Epub 2010 Jan 29. PMID 20226949
- [Background] McGehee DV, Raby M, Carney C, Lee JD, Reyes ML. Extending parental mentoring using an event-triggered video intervention in rural teen drivers. J Safety Res. 2007;38(2):215-27. doi: 10.1016/j.jsr.2007.02.009. Epub 2007 Mar 28. PMID 17478192
- [Background] McCartt AT, Farmer CM, Jenness JW. Perceptions and experiences of participants in a study of in-vehicle monitoring of teenage drivers. Traffic Inj Prev. 2010 Aug;11(4):361-70. doi: 10.1080/15389588.2010.486428. PMID 20730683
- [Background] Curry AE, Peek-Asa C, Hamann CJ, Mirman JH. Effectiveness of Parent-Focused Interventions to Increase Teen Driver Safety: A Critical Review. J Adolesc Health. 2015 Jul;57(1 Suppl):S6-14. doi: 10.1016/j.jadohealth.2015.01.003. PMID 26112737
- [Background] Farah H, Musicant O, Shimshoni Y, Toledo T, Grimberg E, Omer H, Lotan T. Can providing feedback on driving behavior and training on parental vigilant care affect male teen drivers and their parents? Accid Anal Prev. 2014 Aug;69:62-70. doi: 10.1016/j.aap.2013.11.005. Epub 2013 Nov 27. PMID 24331278
- [Derived] Yang J, Peek-Asa C, Zhang Y, Hamann C, Zhu M, Wang Y, Kaur A, Recker R, Rose D, Roth L. ProjectDRIVE: study protocol for a randomized controlled trial to improve driving practices of high-risk teen drivers with a traffic violation. Inj Epidemiol. 2024 Mar 29;11(1):12. doi: 10.1186/s40621-024-00494-5. PMID 38553746